CLINICAL TRIAL: NCT07179185
Title: PRECISE-ECG: Prospective Randomized Evaluation of Clinical Intelligence Support to Reduce Errors in Normal ECGs
Brief Title: Evaluation of Clinical Intelligence Support to Reduce Errors in Normal ECGs
Acronym: PRECISE-ECG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Antonio Luiz Pinho Ribeiro, Full Professor, Internal Medicine Department, School of Medicine, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 409604/2022-4
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Electrocardiogram; Cardiovascular Abnormalities
Keywords: artificial intelligence; electrocardiography; diagnostic methods; telemedicine; normal electrocardiogram
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Specialist Interpretation Without AI (Active Comparator): Specialist physicians interpret normal ECGs without the assistance of the AI-ECG tool. ECGs are routine tracings performed by the Rede de Telemedicina de Minas Gerais (RTMG). Final classification for study endpoints will be based on a panel review by three specialists.
  Interventions: Diagnostic Test: Specialist ECG Interpretation Without AI
- Specialist interpretation with AI assistance (Experimental): Specialist physicians interpret ECGs using the AI-ECG tool, which provides automated classification support indicating whether the ECG is normal or not. ECGs are routine tracings performed by RTMG. Final classification for study endpoints will be based on a panel review by three specialists.
  Interventions: Diagnostic Test: AI-Assisted ECG Interpretation (AI-ECG)

INTERVENTIONS:
Diagnostic Test: AI-Assisted ECG Interpretation (AI-ECG) — Neural network-based AI software that analyzes ECG tracings and provides a classification as normal suggestion to the interpreting specialist.
  Arms: Specialist interpretation with AI assistance
Diagnostic Test: Specialist ECG Interpretation Without AI — Manual interpretation of ECGs by specialists without AI support, following standard diagnostic procedures
  Arms: Control - Specialist Interpretation Without AI

SUMMARY:
This study will evaluate the performance of specialist physicians in interpreting normal electrocardiograms (ECGs) with and without the assistance of an artificial intelligence (AI) neural network. The primary aim is to determine whether AI support affects the rate of false-positive interpretations of normal tracings. Secondary aims include evaluating the time required for interpretation, the sensitivity for detecting abnormalities, and the effect on false positives in ECGs with major abnormalities according to the Minnesota Code system. All ECGs in the sample will be reviewed by a panel of three specialists, to determine the reference classification.

ELIGIBILITY:
Inclusion Criteria:

* ECGs performed routinely by the Rede de Telemedicina de Minas Gerais (RTMG)

Exclusion Criteria:

* ECGs from patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Precision (Positive Predictive Value) for detection of normal ECG tracings | One week
  Precision (Positive Predictive Value) of detecting normal ECG by the physician or physician+model compared against the reference standard defined by a panel of three specialists. Precision (Positive Predictive Value) is defined by the number of true positive normal cases divided by all positive predictions.

SECONDARY OUTCOMES:
Sensitivity, Specificity, Negative Predictive Value, and F1 score for detection of normal ECG tracings | One week
  Accuracy evaluated by Sensitivity, Specificity, Negative Predictive Value, and F1 score of normal ECGs correctly identified by the physician or physician+model, in relation to a reference standard defined by a panel of three specialists.
ECGs with major abnormalities incorrectly classified as normal | One week
  Ratio of ECGs with major abnormalities according to the Minnesota Code system among those incorrectly classified as normal by the physician or physician+model, in relation to a reference standard defined by a panel of three specialists.
Time of analysis for normal cases (seconds per case) | One week
  Time required by the physician, or physician+model, to interpret normal ECGs, measured in seconds per case; the reference standard of normal cases defined by a panel of three specialists.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliveira CRA, Paixao GMM, Tostes VC, Gomes PR, Mendes MS, Paixao MC, Marcolino MS, Ribeiro ALP. Upscaling a regional telecardiology service to a nationwide coverage and beyond: the experience of the Telehealth Network of Minas Gerais. BMJ Glob Health. 2025 Jan 19;10(1):e016692. doi: 10.1136/bmjgh-2024-016692. PMID 39828428
- [Background] Ribeiro ALP, Paixao GMM, Gomes PR, Ribeiro MH, Ribeiro AH, Canazart JA, Oliveira DM, Ferreira MP, Lima EM, Moraes JL, Castro N, Ribeiro LB, Macfarlane PW. Tele-electrocardiography and bigdata: The CODE (Clinical Outcomes in Digital Electrocardiography) study. J Electrocardiol. 2019 Nov-Dec;57S:S75-S78. doi: 10.1016/j.jelectrocard.2019.09.008. Epub 2019 Sep 7. PMID 31526573
- [Background] Ribeiro AH, Ribeiro MH, Paixao GMM, Oliveira DM, Gomes PR, Canazart JA, Ferreira MPS, Andersson CR, Macfarlane PW, Meira W Jr, Schon TB, Ribeiro ALP. Automatic diagnosis of the 12-lead ECG using a deep neural network. Nat Commun. 2020 Apr 9;11(1):1760. doi: 10.1038/s41467-020-15432-4. PMID 32273514